CLINICAL TRIAL: NCT02911818
Title: Combining Lifestyle Modification and Liraglutide to Improve Weight Loss and Health Outcomes
Brief Title: Lifestyle Modification and Liraglutide
Acronym: MODEL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 824806
Record Dates: First submitted 2016-09-06; First posted 2016-09-22 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Liraglutide; Phentermine

STUDY DESIGN:
Masking Description: In the 12 week extension study, participants who are eligible will continue to take liraglutide 3.0 mg in an open fashion. Participants will be randomly assigned in a double-blind fashion to placebo or phentermine.

ARMS (5):
- CMS-Alone (Active Comparator): Lifestyle counseling, as currently recommended by the CMS.
  Interventions: Behavioral: CMS-recommended lifestyle counseling
- CMS-Liraglutide (Active Comparator): CMS lifestyle counselling plus liraglutide.
  Interventions: Behavioral: CMS-recommended lifestyle counseling; Drug: Liraglutide 3.0mg
- Multi-Component Intervention (Active Comparator): CMS-Liraglutide plus a 1000-1200 kcal/day portion-controlled diet prescribed for 12 weeks.
  Interventions: Behavioral: CMS-recommended lifestyle counseling; Drug: Liraglutide 3.0mg; Other: Portion-Controlled Diet
- 12-Week Extension Study: Phentermine Group (Active Comparator): After the 1-year trial, half the participants who join the extension study will be randomized to phentermine 15.0 mg/d in a double-blind fashion, while continuing to take liraglutide. They will also continue to receive monthly lifestyle counseling. To be eligible for the extension study, participants must have been assigned to one of two medication groups in the original study.
  Interventions: Drug: Liraglutide 3.0mg; Drug: Phentermine 15 MG; Behavioral: Extension Study CMS-recommended lifestyle counseling
- 12-Week Extension Study: Placebo Group (Active Comparator): After the 1-year trial, half the participants who join the extension study will be randomized to placebo in a double-blind fashion, while continuing to take liraglutide. They will also continue to receive monthly lifestyle counseling. To be eligible for the extension study, participants must have been assigned to one of two medication groups in the original study.
  Interventions: Drug: Liraglutide 3.0mg; Drug: Placebo Oral Tablet; Behavioral: Extension Study CMS-recommended lifestyle counseling

INTERVENTIONS:
Behavioral: CMS-recommended lifestyle counseling — 21 brief (15 minute) lifestyle counseling visits provided by a physician, nurse practitioner, or registered dietitian.
  Arms: CMS-Alone; CMS-Liraglutide; Multi-Component Intervention
Drug: Liraglutide 3.0mg — Liraglutide is a once-daily self-administered, subcutaneous (beneath the skin) injection.
  Other Names: Saxenda
  Arms: 12-Week Extension Study: Phentermine Group; 12-Week Extension Study: Placebo Group; CMS-Liraglutide; Multi-Component Intervention
Other: Portion-Controlled Diet — A 1000-1200 kcal/day portion-controlled diet prescribed for 12 weeks.
  Arms: Multi-Component Intervention
Drug: Placebo Oral Tablet
  Arms: 12-Week Extension Study: Placebo Group
Drug: Phentermine 15 MG
  Arms: 12-Week Extension Study: Phentermine Group
Behavioral: Extension Study CMS-recommended lifestyle counseling — 4 brief (15 minute) lifestyle counseling visits provided by a physician, nurse practitioner, or registered dietitian.
  Arms: 12-Week Extension Study: Phentermine Group; 12-Week Extension Study: Placebo Group

SUMMARY:
This is a 52 week, single center, open-labeled, randomized controlled trial.

A total of 150 subjects with obesity, who are free of types 1 and 2 diabetes, as well as contraindications to weight loss, will be randomly assigned to one of three treatment groups: 1) lifestyle counseling, as currently recommended by the Centers for Medicare and Medicaid Services (CMS) (i.e., CMS-Alone); 2) CMS lifestyle counseling plus liraglutide (i.e., CMS-Liraglutide); or 3) CMS-Liraglutide plus a portion-controlled diet (i.e., Multi-Component Intervention).

Subjects in all three groups will have 14 brief (15 minute) lifestyle counseling visits the first 24 weeks, followed by monthly visits in weeks 25-52. This is the schedule and duration of counseling visits recommended by CMS. Counseling sessions will be delivered by a physician, nurse practitioner or registered dietitian (RD) working in consultation with the former providers.

Subjects in all three groups also will have brief physician visits at weeks 1, 4, 8, 16, 24, 36, and 52 (total of 7 visits). These visits are needed for subjects in both liraglutide groups to monitor their response to the medication. These visits are included for subjects in CMS-Alone to match the intensity of medical care provided the two other groups.

The primary outcome is % reduction in initial body weight, as measured from randomization to week 52. Secondary outcomes include the proportion of participants who at week 52 lose >5%, >10%, and >15% of initial weight, as well as % reduction in weight at week 24 and the proportion of participants who meet the three categorical weight losses at this time. The secondary efficacy measures include changes (from randomization to week 52) in cardiovascular disease (CVD) risk factors, glycemic control, mood, quality of life, eating behavior, appetite, sleep, and satisfaction with weight loss.

Safety endpoints will include physical examination, adverse events (AEs), standard laboratory tests, and mental health assessed by the Columbia Suicidality Severity Rating Scale (C-SSRS) and Patient Health Questionnaire (PHQ-9).

Statistical Analysis. Using a sample size equation for longitudinal clustered samples, a randomization sample of 50 subjects in CMS-Alone, 50 in CMS-Liraglutide, and 50 in the Multi-Component Intervention provides >80% power to detect the two primary contrasts to be statistically significant. This estimate allows for 20% attrition during the 52-week trial, resulting in approximately 40 treatment completers per group. The ITT longitudinal statistical design will further improve power by allowing the inclusion of available data for non-completers and the adjustment of possible variance reducing baseline covariates.

DETAILED DESCRIPTION:
The addendum to the original 52-week trial, is a 12-week, single center, randomized placebo-controlled, parallel group designed trial. This 12-week extension study is separate from the original 52-week trial and will not affect the outcome or analysis of the 52-week, 3-arm trial.

Participants and investigators will be masked to participants' assignment to phentermine 15 mg/d versus placebo. Participants in both groups will receive liraglutide in an open-label manner.

We anticipate that 23 (of 50) participants from the original CMS-Liraglutide group and 23 (of 50) from the Multi-Component Intervention will be eligible to participate in the extension study and will elect to do so. We anticipate that 20 participants in each group will complete the 12-week extension study and that those who receive liraglutide 3.0 mg plus phentermine 15.0 mg/d will lose, from randomization to week 12, 3.5+3.5% of initial weight, compared with 0.0+0.5% for those assigned to liraglutide plus placebo.

All participants in the extension study will meet with a physician or nurse practitioner at randomization (week 0) and at weeks 2, 4, 8 and 12. On each occasion they will review patients' blood pressure and pulse, assess suicidal ideation, and record and respond appropriately to reports of changes in physical health. As during the 1-year prior trial, brief lifestyle counseling (15 min) will provided at monthly visits (excluding week 2) by the physician or nurse practitioner or by a registered dietitian or behavioral psychologist, working under their supervision. The lifestyle intervention will be the same as that provided during the last 6 months of both the CMS-Liraglutide and Multi-Component interventions.

Following the 12-week randomized trial, phentermine (or placebo) will be terminated, and all participants will continue to receive liraglutide 3.0 mg/d for an additional 8 weeks (i.e., weeks 12-20) and have lifestyle counseling and medical assessments at weeks 16 and 20. Liraglutide 3.0 mg/d will be terminated at week 20, and participants will have a final safety assessment at week 24.

The primary endpoint of the 12-week extension trial is change in body weight (i.e., % reduction in randomization weight), as measured from randomization (week 0) to week 12. Secondary endpoints include the proportion of subjects who lose > 5% or > 10% of initial weight from randomization to week 12, as well as changes from randomization to week 12 in cardiovascular disease (CVD) risk factors (i.e, blood pressure, triglycerides, LDL and HDL cholesterol, and waist circumference), glycemic control (i.e., fasting blood sugar), mood (PHQ-9), quality of life (i.e, SF-36 and IWQOL-Lite), eating behavior (i.e., Eating Inventory, Eating Disorder Examination-Questionnaire, and Yale Food Addiction Scale), appetite (i.e., visual analogue scales), sleep (i.e., Pittsburgh Sleep Quality Index), and weight loss satisfaction. (All of these measures were administered in the original 1-year trial.)

Safety endpoints will include physical examination, adverse events (AEs), standard laboratory tests, and mental health assessed by the Columbia Suicidality Severity Rating Scale (C-SSRS) and Patient Health Questionnaire (PHQ-9).

All data analyses will proceed using the same principles and methods used in the original protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have a BMI ≥ 30 and ≤ 55 kg/m²
2. Age ≥ 21 years and ≤ 70 years
3. Eligible female patients will be:

   * non-pregnant, evidenced by a negative urine dipstick pregnancy test
   * non-lactating
   * surgically sterile or postmenopausal, or they will agree to continue to use an accepted method of birth control during the study
4. Ability to provide informed consent before any trial-related activities
5. Participants must:

   * have a primary care provider (PCP) who is responsible for providing routine care
   * have a reliable telephone service with which to communicate with study staff
   * understand and be willing to comply with all study-related procedures and agree to participate in the study by giving written informed consent
   * plan to remain in the Philadelphia area for the next 18 months

Exclusion Criteria:

1. Pregnant or nursing, or plans to become pregnant in the next 18 months, or not using adequate contraceptive measures
2. Personal or family history of medullary thyroid cancer or multiple endocrine neoplasia syndrome type 2
3. Uncontrolled hypertension (systolic blood pressure ≥ 160 mm Hg or diastolic blood pressure ≥ 100 mm Hg)
4. Type 1 diabetes
5. Type 2 diabetes
6. A fasting glucose ≥ 126 mg/dl (on second assessment after first elevated value)
7. Recent history of cardiovascular disease (e.g., myocardial infarction or stroke within the past 6 months), congestive heart failure, or heart block greater than first degree
8. Clinically significant hepatic or renal disease
9. Thyroid disease, not controlled
10. History of malignancy (except for non-melanoma skin cancer) in past 5 years
11. Current major depressive episode, active suicidal ideation, or history of suicide attempts
12. Psychiatric hospitalization within the past 6 months
13. Self-reported alcohol or substance abuse within the past 12 months, including at-risk drinking (current consumption of ≥ 14 alcoholic drinks per week)
14. Use in past 3 months of medications known to induce significant weight loss (i.e., prescription weight loss medications) or weight gain (e.g., chronic use of oral steroids, second generation antipsychotics)
15. Loss of ≥ 10 lb of body weight within the past 3 months
16. History of (or plans for) bariatric surgery
17. Inability to walk 5 blocks comfortably or engage in some other form of aerobic activity (e.g., swimming)
18. Known or suspected allergy to trial medication(s), excipients, or related products
19. Hypersensitivity to liraglutide or any product components
20. The receipt of any investigational drug within 6 months prior to this trial
21. Previous participation in this trial (e.g., randomized and failed to participate)
22. History of pancreatitis
23. Subjects will be included/excluded according to the latest updated US PI.

12-Week Extension Trial:

Inclusion Criteria

Inclusion criteria are those described for the original 1-year trial (enumerated above). The principal exception from these criteria is that participants will only be required to have a BMI > 27 kg/m2, with or without co-morbidities, to be eligible to participate in the extension study. All participants will have met BMI inclusion criteria when they initiated the use of liraglutide and now will use it, potentially with phentermine 15 mg/d, to facilitate to the maintenance of lost weight. (Liraglutide is approved for chronic weight management, including following successful weight loss.) We do not wish to enroll participants with a BMI < 27 kg/m2 because of the possibility that they could reduce substantially below a BMI of 24.9 kg/m2, the upper limit of "normal" weight.

Exclusion Criteria:

Exclusion criteria will include those listed in the original protocol, including those specific to the use of liraglutide 3.0 mg/d (e.g., family history of medullary thyroid cancer).

Additional exclusion criteria added to the 12-week extension study are specific to the use of phentermine 15 mg/d. They include:

1. Use of monoamine oxidase inhibitors in the past 2 weeks
2. Glaucoma
3. Presence or history of marked agitation
4. History of drug abuse
5. Known hypersensitivity to sympathomimetic amines
6. Current use of selective serotonin re-uptake inhibitors (e.g., fluoxetine, sertraline, etc)
7. Current use of any other weight loss medications (besides liraglutide 3.0 mg/d)
8. History of coronary artery disease

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Wadden, Ph.D., Principal Investigator — University of Pennsylvania, Center for Weight and Eating Disorders
Locations (1):
- University of Pennsylvania Center for Weight and Eating Disorders, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tronieri JS, Wadden TA, Walsh O, Berkowitz RI, Alamuddin N, Gruber K, Leonard S, Bakizada ZM, Chao AM. Effects of liraglutide on appetite, food preoccupation, and food liking: results of a randomized controlled trial. Int J Obes (Lond). 2020 Feb;44(2):353-361. doi: 10.1038/s41366-019-0348-6. Epub 2019 Mar 29. PMID 30926955
- [Derived] Tronieri JS, Wadden TA, Walsh OA, Berkowitz RI, Alamuddin N, Gruber K, Leonard S, Chao AM. Effects of liraglutide plus phentermine in adults with obesity following 1 year of treatment by liraglutide alone: A randomized placebo-controlled pilot trial. Metabolism. 2019 Jul;96:83-91. doi: 10.1016/j.metabol.2019.03.005. Epub 2019 Mar 20. PMID 30902750
- [Derived] Wadden TA, Walsh OA, Berkowitz RI, Chao AM, Alamuddin N, Gruber K, Leonard S, Mugler K, Bakizada Z, Tronieri JS. Intensive Behavioral Therapy for Obesity Combined with Liraglutide 3.0 mg: A Randomized Controlled Trial. Obesity (Silver Spring). 2019 Jan;27(1):75-86. doi: 10.1002/oby.22359. Epub 2018 Nov 13. PMID 30421856
- See also: Center for Weight and Eating Disorders Website — https://www.med.upenn.edu/weight/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial enrolled 150 participants for the original 52-week study. The 12-week extension study randomized 45 participants from the 100 eligible from the original 52-week trial who were originally in either the CMS-Liraglutide or Multi-Component groups. Eligible participants for the 12-week extension had to complete 1 year on liraglutide.
Groups:
- CMS-Alone: Lifestyle counseling on the visit schedule recommended by the Centers for Medicare and Medicaid Services (CMS).
  CMS-recommended lifestyle counseling: 21 brief (15 minute) lifestyle counseling visits provided by a physician, nurse practitioner, or registered dietitian.
- CMS-Liraglutide: CMS lifestyle counselling plus liraglutide 3.0 mg/d.
  CMS-recommended lifestyle counseling: 21 brief (15 minute) lifestyle counseling visits provided by a physician, nurse practitioner, or registered dietitian.
  Liraglutide 3.0mg/d: Liraglutide is a once-daily self-administered, subcutaneous (beneath the skin) injection.
- Multi-Component Intervention: CMS-Liraglutide plus a 1000-1200 kcal/day portion-controlled diet.
  CMS-recommended lifestyle counseling: 21 brief (15 minute) lifestyle counseling visits provided by a physician, nurse practitioner, or registered dietitian.
  Liraglutide 3.0mg/d: Liraglutide is a once-daily self-administered, subcutaneous (beneath the skin) injection.
  Portion-Controlled Diet: A 1000-1200 kcal/day portion-controlled diet prescribed for 12 weeks, beginning at week 4.
- 12-Week Extension Study: Phentermine Group: After the 1-year trial, half the participants who elect to join the extension study will be randomized to phentermine 15.0 mg/d in a double-blind fashion, while continuing to take liraglutide. They will also continue to receive monthly lifestyle counseling: 4 brief (15 minute) lifestyle counseling visits provided by a physician, nurse practitioner, or registered dietitian.
  Liraglutide 3.0mg/d: Liraglutide is a once-daily self-administered, subcutaneous (beneath the skin) injection.
  Phentermine 15 MG
- 12-Week Extension Study: Placebo Group: After the 1-year trial, half the participants who elect to join the extension study will be randomized to placebo in a double-blind fashion, while continuing to take liraglutide. They will also continue to receive monthly lifestyle counseling: 4 brief (15 minute) lifestyle counseling visits provided by a physician, nurse practitioner, or registered dietitian.
  Liraglutide 3.0mg/d: Liraglutide is a once-daily self-administered, subcutaneous (beneath the skin) injection.
  Placebo Oral Tablet
Period: 52 Week Study
Arm/Group | CMS-Alone | CMS-Liraglutide | Multi-Component Intervention | 12-Week Extension Study: Phentermine Group | 12-Week Extension Study: Placebo Group
Started | 50 | 50 | 50 | 0 | 0
Completed | 46 | 45 | 46 | 0 | 0
Not Completed | 4 | 5 | 4 | 0 | 0
Period: 12 Week Extension Study
Arm/Group | CMS-Alone | CMS-Liraglutide | Multi-Component Intervention | 12-Week Extension Study: Phentermine Group | 12-Week Extension Study: Placebo Group
Started | 0 | 0 | 0 | 22 | 23
Completed | 0 | 0 | 0 | 22 | 22
Not Completed | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- CMS-Alone: Lifestyle counseling, on the visit schedule currently recommended by the CMS.
  CMS-recommended lifestyle counseling: 21 brief (15 minute) lifestyle counseling visits provided by a physician, nurse practitioner, or registered dietitian.
- Total: Total of all reporting groups
Arm/Group | CMS-Alone | CMS-Liraglutide | Multi-Component Intervention | Total
Number analyzed (Participants) | 50 | 50 | 50 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (11.0) | 45.2 (12.3) | 48.0 (11.9) | 47.6 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 42 | 38 | 119
  Male | 11 | 8 | 12 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 22 | 23 | 22 | 67
  White | 27 | 27 | 27 | 81
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Baseline Weight
Time Frame: Randomization and 52 weeks
Measure: Mean (Standard Error); unit: percent change
Arm/Group | CMS-Alone | CMS-Liraglutide | Multi-Component Intervention
Number analyzed (Participants) | 50 | 50 | 50
percent change | -6.1 (1.3) | -11.5 (1.3) | -11.8 (1.3)

2. Primary Outcome: Extension Study Primary Outcome: Percent Change in Re-randomization Weight
Time Frame: Re-randomization and 12 weeks
Measure: Mean (Standard Error); unit: percent change
Arm/Group | 12-Week Extension Study: Phentermine Group | 12-Week Extension Study: Placebo Group
Number analyzed (Participants) | 22 | 23
percent change | -1.6 (0.6) | -0.1 (0.5)

3. Secondary Outcome: Change in Systolic Blood Pressure
Time Frame: Randomization and 52 weeks
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | CMS-Alone | CMS-Liraglutide | Multi-Component Intervention
Number analyzed (Participants) | 50 | 50 | 50
mm Hg | -14.1 (2.1) | -13.3 (2.1) | -15.3 (2.1)

4. Secondary Outcome: Change in Diastolic Blood Pressure
Time Frame: Randomization and 52 weeks
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | CMS-Alone | CMS-Liraglutide | Multi-Component Intervention
Number analyzed (Participants) | 50 | 50 | 50
mm Hg | -3.0 (1.2) | -2.9 (1.2) | -3.5 (1.2)

5. Secondary Outcome: Change in Heart Rate
Time Frame: Randomization and 52 weeks
Measure: Mean (Standard Error); unit: Beats per minute
Arm/Group | CMS-Alone | CMS-Liraglutide | Multi-Component Intervention
Number analyzed (Participants) | 50 | 50 | 50
Beats per minute | -7.4 (2.0) | -5.3 (2.0) | 9.7 (2.0)

6. Secondary Outcome: Change in Waist Circumference
Time Frame: Randomization and 52 weeks
Measure: Mean (Standard Error); unit: cm
Arm/Group | CMS-Alone | CMS-Liraglutide | Multi-Component Intervention
Number analyzed (Participants) | 50 | 50 | 50
cm | -6.5 (1.3) | -11.1 (1.3) | -12.6 (1.3)

7. Secondary Outcome: Change in Total Cholesterol
Time Frame: Randomization and 52 weeks
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | CMS-Alone | CMS-Liraglutide | Multi-Component Intervention
Number analyzed (Participants) | 50 | 50 | 50
mg/dL | -7.0 (3.5) | -9.7 (3.6) | -10.0 (3.5)

8. Secondary Outcome: Change in LDL Cholesterol
Time Frame: Randomization and 52 weeks
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | CMS-Alone | CMS-Liraglutide | Multi-Component Intervention
Number analyzed (Participants) | 50 | 50 | 50
mg/dL | -3.3 (3.1) | -9.6 (3.1) | -9.4 (3.1)

9. Secondary Outcome: Change in HDL Cholesterol
Time Frame: Randomization and 52 weeks
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | CMS-Alone | CMS-Liraglutide | Multi-Component Intervention
Number analyzed (Participants) | 50 | 50 | 50
mg/dL | -1.3 (1.3) | 3.0 (1.3) | 2.0 (1.3)

10. Secondary Outcome: Change in Triglycerides
Time Frame: Randomization and 52 weeks
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | CMS-Alone | CMS-Liraglutide | Multi-Component Intervention
Number analyzed (Participants) | 50 | 50 | 50
mg/dL | -16.3 (5.7) | -21.3 (5.8) | -14.4 (5.7)

11. Secondary Outcome: Change in C Reactive Protein
Time Frame: Randomization and 52 weeks
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | CMS-Alone | CMS-Liraglutide | Multi-Component Intervention
Number analyzed (Participants) | 50 | 50 | 50
mg/L | -0.4 (0.7) | -2.0 (0.7) | -3.0 (0.7)

12. Secondary Outcome: Change in Fasting Glucose
Time Frame: Randomization and 52 weeks
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | CMS-Alone | CMS-Liraglutide | Multi-Component Intervention
Number analyzed (Participants) | 50 | 50 | 50
mg/dL | 0.01 (1.3) | -5.2 (1.3) | -5.7 (1.3)

13. Secondary Outcome: Change in HbA1c
Time Frame: Randomization and 52 weeks
Measure: Mean (Standard Error); unit: percentage
Arm/Group | CMS-Alone | CMS-Liraglutide | Multi-Component Intervention
Number analyzed (Participants) | 50 | 50 | 50
percentage | -0.3 (0.03) | -0.5 (0.03) | -0.6 (0.03)

14. Secondary Outcome: Change in Fasting Insulin
Time Frame: Randomization and 52 weeks
Measure: Mean (Standard Error); unit: uIU/mL
Arm/Group | CMS-Alone | CMS-Liraglutide | Multi-Component Intervention
Number analyzed (Participants) | 50 | 50 | 50
uIU/mL | -1.5 (0.8) | -1.1 (0.8) | -1.5 (0.8)

15. Secondary Outcome: Change in HOMA-IR
Description: HOMA-IR is a measurement for insulin resistance and is calculated from: fasting insulin (U/L) x fasting glucose (mg/dL)/405. A decrease from baseline to the end of treatment, a negative value, indicates an improvement
Time Frame: Randomization and 52 weeks
Measure: Mean (Standard Error); unit: mg/dL*µIU/mL/405
Arm/Group | CMS-Alone | CMS-Liraglutide | Multi-Component Intervention
Number analyzed (Participants) | 50 | 50 | 50
mg/dL*µIU/mL/405 | -0.4 (0.2) | -0.3 (0.2) | -0.4 (0.2)

16. Secondary Outcome: Change in 36-Item Short Form Survey (SF-36) - Physical Component Summary
Description: All sub scales are scored from 0 - 100, with higher scores indicating better health. Each component summary is a normed score with a mean of 50 and standard deviation of 10 in the US general population. Higher scores indicate better health.
  Z-scores are computed for each subscale, which are then converted into a component summary z-score using a weighted formula. The component summary z-score is then converted to a t-distribution with a mean of 50 and standard deviation of 10.
  Scores are scaled to a T-score with a mean of 50 and standard deviation of 10. Scores above 50 indicate better health.
Time Frame: Randomization and 52 weeks
Measure: Mean (Standard Error); unit: T scores
Arm/Group | CMS-Alone | CMS-Liraglutide | Multi-Component Intervention
Number analyzed (Participants) | 50 | 50 | 50
T scores | 4.4 (1.0) | 2.1 (1.0) | 3.4 (1.0)

17. Secondary Outcome: Change 36-Item Short Form Survey (SF-36) - Mental Component Summary
Description: as for outcome 16
Time Frame: Randomization and 52 weeks
Measure: Mean (Standard Error); unit: T scores
Arm/Group | CMS-Alone | CMS-Liraglutide | Multi-Component Intervention
Number analyzed (Participants) | 50 | 50 | 50
T scores | 0.8 (1.3) | 4.5 (1.3) | 6.4 (1.3)

18. Secondary Outcome: Change in Patient Health Questionnaire (PHQ-9)
Description: PHQ-9 is scored based on a 0-27 scale in which higher scores indicate more severe depression. Values are summed to compute the total score.
Time Frame: Randomization and 52 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CMS-Alone | CMS-Liraglutide | Multi-Component Intervention
Number analyzed (Participants) | 50 | 50 | 50
score on a scale | -1.8 (0.6) | -1.9 (0.6) | -1.5 (0.6)

19. Secondary Outcome: Extension Study Secondary Outcome: Change in Systolic Blood Pressure
Time Frame: Re-randomization and 12 weeks
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | 12-Week Extension Study: Placebo Group | 12-Week Extension Study: Phentermine Group
Number analyzed (Participants) | 23 | 22
mm Hg | 1.2 (2.1) | 2.0 (2.1)

20. Secondary Outcome: Extension Study Secondary Outcome: Change in Diastolic Blood Pressure
Time Frame: Re-randomization and 12 weeks
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | 12-Week Extension Study: Phentermine Group | 12-Week Extension Study: Placebo Group
Number analyzed (Participants) | 22 | 23
mm Hg | 1.3 (1.6) | 0.2 (1.6)

21. Secondary Outcome: Extension Study Secondary Outcome: Change in Heart Rate
Time Frame: Re-randomization and 12 weeks
Measure: Mean (Standard Error); unit: Beats per minute
Arm/Group | 12-Week Extension Study: Placebo Group | 12-Week Extension Study: Phentermine Group
Number analyzed (Participants) | 23 | 22
Beats per minute | 0 (1.4) | 2.1 (1.4)

22. Secondary Outcome: Extension Study Secondary Outcome: Change in Waist Circumference
Time Frame: Re-randomization and 12 weeks
Measure: Mean (Standard Error); unit: cm
Arm/Group | 12-Week Extension Study: Placebo Group | 12-Week Extension Study: Phentermine Group
Number analyzed (Participants) | 23 | 22
cm | -0.6 (0.8) | -0.4 (0.8)

23. Secondary Outcome: Extension Study Secondary Outcome: Change in Total Cholesterol
Time Frame: Re-randomization and 12 weeks
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | 12-Week Extension Study: Placebo Group | 12-Week Extension Study: Phentermine Group
Number analyzed (Participants) | 23 | 22
mg/dL | 3.4 (3.3) | 0.4 (3.3)

24. Secondary Outcome: Extension Study Secondary Outcome: Change in LDL Cholesterol
Time Frame: Re-randomization and 12 weeks
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | 12-Week Extension Study: Placebo Group | 12-Week Extension Study: Phentermine Group
Number analyzed (Participants) | 23 | 22
mg/dL | 2.3 (2.8) | -2.4 (2.8)

25. Secondary Outcome: Extension Study Secondary Outcome: Change in HDL Cholesterol
Time Frame: Re-randomization and 12 weeks
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | 12-Week Extension Study: Placebo Group | 12-Week Extension Study: Phentermine Group
Number analyzed (Participants) | 23 | 22
mg/dL | 0.6 (1.4) | 2.0 (1.4)

26. Secondary Outcome: Extension Study Secondary Outcome: Change in Triglycerides
Time Frame: Re-randomization and 12 weeks
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | 12-Week Extension Study: Placebo Group | 12-Week Extension Study: Phentermine Group
Number analyzed (Participants) | 23 | 22
mg/dL | 4.1 (4.7) | 6.6 (4.7)

27. Secondary Outcome: Extension Study Secondary Outcome: Change in c-Reactive Protein
Time Frame: Re-randomization and 12 weeks
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | 12-Week Extension Study: Placebo Group | 12-Week Extension Study: Phentermine Group
Number analyzed (Participants) | 23 | 22
mg/L | -0.8 (0.6) | -0.6 (0.6)

28. Secondary Outcome: Extension Study Secondary Outcome: Change in Fasting Glucose
Time Frame: Re-randomization and 12 weeks
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | 12-Week Extension Study: Placebo Group | 12-Week Extension Study: Phentermine Group
Number analyzed (Participants) | 23 | 22
mg/dL | 1.4 (1.6) | 6.3 (1.6)

29. Secondary Outcome: Extension Study Secondary Outcome: Change in HbA1c
Time Frame: Re-randomization and 12 weeks
Measure: Mean (Standard Error); unit: percentage
Arm/Group | 12-Week Extension Study: Placebo Group | 12-Week Extension Study: Phentermine Group
Number analyzed (Participants) | 23 | 22
percentage | 0.0 (0.1) | 0.0 (0.0)

30. Secondary Outcome: Extension Study Secondary Outcome: Change in Fasting Insulin
Time Frame: Re-randomization and 12 weeks
Measure: Mean (Standard Error); unit: uIU/mL
Arm/Group | 12-Week Extension Study: Placebo Group | 12-Week Extension Study: Phentermine Group
Number analyzed (Participants) | 23 | 22
uIU/mL | 0.2 (1.0) | 0.5 (1.0)

31. Secondary Outcome: Extension Study Secondary Outcome: Change in HOMA-IR
Description: as for outcome 15
Time Frame: Re-randomization and 12 weeks
Measure: Mean (Standard Error); unit: mg/dL*µIU/mL/405
Arm/Group | 12-Week Extension Study: Placebo Group | 12-Week Extension Study: Phentermine Group
Number analyzed (Participants) | 23 | 22
mg/dL*µIU/mL/405 | 0.1 (0.2) | 0.3 (0.2)

32. Secondary Outcome: Extension Study Secondary Outcome: SF-36 - Physical Health Component
Description: as for outcome 16
Time Frame: Re-randomization and 12 weeks
Measure: Mean (Standard Error); unit: T scores
Arm/Group | 12-Week Extension Study: Placebo Group | 12-Week Extension Study: Phentermine Group
Number analyzed (Participants) | 23 | 22
T scores | 0.3 (1.0) | -1.2 (1.0)

33. Secondary Outcome: Extension Study Secondary Outcome: SF-36 - Mental Health Component
Description: as for outcome 16
Time Frame: Re-randomization and 12 weeks
Measure: Mean (Standard Error); unit: T scores
Arm/Group | 12-Week Extension Study: Placebo Group | 12-Week Extension Study: Phentermine Group
Number analyzed (Participants) | 23 | 22
T scores | -0.1 (1.1) | 0.2 (1.1)

34. Secondary Outcome: Extension Study Secondary Outcome: Patient Health Questionnaire (PHQ-9)
Description: as for outcome 18
Time Frame: Re-randomization and 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 12-Week Extension Study: Placebo Group | 12-Week Extension Study: Phentermine Group
Number analyzed (Participants) | 23 | 22
score on a scale | 0.2 (0.4) | 0.0 (0.4)

ADVERSE EVENTS:
Time Frame: 52-weeks post randomization for the original trial; 12-weeks for the extension trial post extension randomization
Groups:
- Multi-Component Intervention: CMS-Liraglutide plus a 1000-1200 kcal/day portion-controlled diet.
  CMS-recommended lifestyle counseling: 21 brief (15 minute) lifestyle counseling visits provided by a physician, nurse practitioner, or registered dietitian.
  Liraglutide 3.0mg: Liraglutide is a once-daily self-administered, subcutaneous (beneath the skin) injection.
  Portion-Controlled Diet: A 1000-1200 kcal/day portion-controlled diet prescribed for 12 weeks, beginning at week 4.
- 12-Week Extension Study: Phentermine Group: After the 1-year trial, half the participants who join the extension study will be randomized to phentermine 15.0 mg/d in a double-blind fashion, while continuing to take liraglutide. They will also continue to receive monthly lifestyle counseling.
  CMS-recommended lifestyle counseling: 4 brief (15 minute) lifestyle counseling visits provided by a physician, nurse practitioner, or registered dietitian.
  Liraglutide 3.0mg: Liraglutide is a once-daily self-administered, subcutaneous (beneath the skin) injection.
  Phentermine 15 MG
- 12-Week Extension Study: Placebo Group: After the 1-year trial, half the participants who join the extension study will be randomized to placebo in a double-blind fashion, while continuing to take liraglutide. They will also continue to receive monthly lifestyle counseling.
  CMS-recommended lifestyle counseling: 4 brief (15 minute) lifestyle counseling visits provided by a physician, nurse practitioner, or registered dietitian.
  Liraglutide 3.0mg: Liraglutide is a once-daily self-administered, subcutaneous (beneath the skin) injection.
  Placebo Oral Tablet
Arm/Group | CMS-Alone | CMS-Liraglutide | Multi-Component Intervention | 12-Week Extension Study: Phentermine Group | 12-Week Extension Study: Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 1/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 2/50 | 0/50 | 3/50 | 1/22 | 0/23
Other Adverse Events (participants affected / at risk) | 21/50 | 42/50 | 44/50 | 12/22 | 11/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CMS-Alone (N=50) | CMS-Liraglutide (N=50) | Multi-Component Intervention (N=50) | 12-Week Extension Study: Phentermine Group (N=22) | 12-Week Extension Study: Placebo Group (N=23)
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Quadriplegic event (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CMS-Alone (N=50) | CMS-Liraglutide (N=50) | Multi-Component Intervention (N=50) | 12-Week Extension Study: Phentermine Group (N=22) | 12-Week Extension Study: Placebo Group (N=23)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 16 (18) | 14 (18) | 1 (1) | 2 (2)
Gastroenteritis (Gastrointestinal disorders) | 2 (2) | 10 (12) | 8 (8) | 2 (2) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Depressed mood (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Tonsillopharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Lower back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Knee pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 4 (4) | 5 (6) | 0 (0) | 0 (0)
Injection site irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 6 (6) | 0 (0) | 0 (0)
Gastroesophageal reflux disorder (Gastrointestinal disorders) | 2 (2) | 2 (2) | 6 (9) | 3 (3) | 1 (1)
Vomitting (Gastrointestinal disorders) | 3 (3) | 6 (8) | 5 (6) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 6 (9) | 7 (7) | 2 (2) | 1 (2)
Musculoskeletal injury (Musculoskeletal and connective tissue disorders) | 6 (7) | 6 (6) | 12 (12) | 1 (1) | 5 (6)
Constipation (Gastrointestinal disorders) | 1 (2) | 15 (16) | 17 (21) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 18 (21) | 13 (17) | 2 (2) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Heart Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Restlessness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/18/NCT02911818/Prot_SAP_000.pdf